CLINICAL TRIAL: NCT02434354
Title: A Phase Ib Tissue Collection Study of Pembrolizumab (MK-3475) in Subjects With Resectable Advanced Melanoma
Brief Title: A Tissue Collection Study of Pembrolizumab (MK-3475) in Subjects With Resectable Advanced Melanoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 01615
Record Dates: First submitted 2015-04-30; First posted 2015-05-05 (Estimated); Results first posted 2021-01-05 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-05

CONDITIONS: Malignant Melanoma
Keywords: Clinical stage III or resectable stage IV melanoma (MEL)
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- neo-adjuvant/adjuvant pembrolizaumab 200 mg IV (Experimental): All subjects will receive 1 cycle neo-adjuvant pembrolizumab 200mg IV followed by complete surgical resection followed by pembrolizumab Q3weeks for 1 year
  Interventions: Drug: pembrolizumab

INTERVENTIONS:
Drug: pembrolizumab — 200 mg Subjects will receive 1 dose of neoadjuvant pembrolizumab, followed by complete resection and then a year of adjuvant pembrolizumab
  Other Names: keytruda

SUMMARY:
The main purpose of this trial is to evaluate the safety, tolerability and adverse event profile of pembrolizumab in subjects who have high risk melanoma before and after their standard of care surgical resection, and to collect tumor tissue from subjects before and after receipt of pembrolizumab to look at how the experimental drug interacts with tumor tissue. Subjects will receive 1 dose of neoadjuvant pembrolizumab, followed by complete resection and then a year of adjuvant pembrolizumab

DETAILED DESCRIPTION:
detailed description listed above

ELIGIBILITY:
Inclusion Criteria:

1. The subject must have clinical stage III or resectable stage IV MEL. Subject's may not have a diagnosis of uveal or mucosal melanoma.
2. The subject must be expected to have an adequate amount of tumor burden to yield 2-4 pre-operative research core biopsy (14-gauge needle) specimens or the equivalent amount of tissue (4-6 mm punch biopsy), in addition, to the tissue required for diagnostic purposes.
3. The subject must be expected to have an adequate amount of residual tumor after their pre-operative research tumor tissue collection, such that their operative research tumor collection will also yield at least 4-6 research core biopsy specimens or the equivalent amount of tissue
4. The subject must be willing to undergo the two paired tumor tissue biopsy procedures to obtain samples for biomarker analysis. Tissue obtained must not be previously irradiated.
5. Either the subject or the subject's legal representative must be willing and able to provide written informed consent for the trial.
6. The subject must be ≥ 18 years of age on day of signing informed consent.
7. The subject must have a performance status of 0 or 1 on the ECOG Performance Scale.
8. The subject must demonstrate adequate organ function as defined in Table 1, all screening labs must be performed within 10 days of treatment initiation.

   Table 1 Adequate Organ Function Laboratory Values System Laboratory Value Hematological Absolute neutrophil count (ANC)
   * 1500/mcL Platelets
   * 100,000/ mcL Hemoglobin
   * 9 g/dL or ≥5.6 mmol/L Renal Serum creatinine OR Measured or calculated creatinine clearance (GFR can also be used in place of creatinine or CrCl)

     ≤1.5 X upper limit of normal (ULN) OR
   * 50 mL/min for subject with creatinine levels > 1.5 X institutional ULN UPCC# 01615: Tissue Collection Study of Pembrolizumab in Advanced Melanoma Version Date: 12/30/2014 Page 10 Hepatic Serum total bilirubin

     * 1.5 X ULN OR Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT)
     * 2.5 X ULN OR
     * 5 X ULN for subjects with liver metastases Coagulation International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT)
     * 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
     * 1.5 X ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants aCreatinine clearance should be calculated per institutional standard.
9. Female subject's of childbearing potential must have a negative serum pregnancy test within 72 hours prior to receiving the first dose of study medication.
10. The subject must be willing to use protocol defined method(s) of contraception:

Female subjects of childbearing potential must be willing to use 2 methods of contraception, or abstain from heterosexual sexual intercourse for two weeks before the time of the first dose of study medication, while on study, through 120 days after the last dose of study medication.

Female subject's of childbearing potential are defined as those women who have not been surgically sterilized or have not been free from menses for > 1 year.

Male subjects must agree to use an adequate method of contraception starting with the first dose of study medication, while on study, through 120 days after the last dose of study medication.

Acceptable forms of birth control include condoms, diaphragms, cervical cap, an intra-uterine device (IUD), surgical sterility (tubal ligation or a partner that has undergone a vasectomy), or oral contraceptives, OR the subject must agree to completely abstain from heterosexual intercourse. Abstinence at certain times of the cycle only, such as during the days of ovulation, after ovulation and withdrawal are not acceptable methods of birth control

Exclusion Criteria:

1. Subject has unresectable disease; i.e. in the opinion of the surgical oncologist, all of the subject's melanoma cannot be completely removed with a clear margin.
2. Subject is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of study treatment.
3. Subject has a known hypersensitivity to pembrolizumab or any of its ingredients.
4. Subject has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to enrollment.
5. Subject has had a prior monoclonal antibody within 4 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
6. Subject has received prior therapy with an anti-PD-1, anti-PD-L1, anti-PD-L2, anti-CD137, or anti-Cytotoxic T-lymphocyte-associated antigen-4 (CTLA-4) agents (including ipilimumab), interferon, high dose IL-1 or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways.
7. Subject has had prior chemotherapy, targeted small molecule therapy, 2 weeks prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion
8. For subject's who have received major surgery, the subject must have recovered adequately from the toxicity and/or complications from the intervention prior to starting study therapy.
9. Subject has had radiation therapy to the tumor selected for research collection, or has had radiation therapy to any site within 4 weeks prior to study Day 1.
10. Subject has received transfusion of blood products (including platelets or red blood cells) or administration of colony stimulating factors (including G-CSF, GM-CSF or recombinant erythropoietin) within 4 weeks prior to study Day 1.
11. Subject has a known additional malignancy that is progressing or requires active treatment.
12. Subject has known active central nervous system (CNS) metastases and/or carcinomatous meningitis.

    Note: Subjects with previously treated brain metastases will be eligible to participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment.
13. Subject has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents.

    Note: Subjects with vitiligo or resolved childhood asthma/atopy are an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections will not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
14. Subject has evidence of interstitial lung disease or active, non-infectious pneumonitis.
15. Subject has an active infection requiring systemic therapy, including active tuberculosis
16. Subject has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
17. Subject has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
18. Subject is pregnant or breastfeeding, or expecting to conceive or father a child within the projected duration of the trial participation (from 2 weeks prior to the first dose of study treatment, while participating on the study and through 120 days after the last dose of trial treatment).
19. Subject has severe cardiovascular disease, i.e. arrhythmias, requiring chronic treatment, congestive heart failure (NYHA Class III or IV) or symptomatic ischemic heart disease.
20. Subject has hepatic decompensation (Child-Pugh score >6 [class B and C]).
21. Subject has uncontrolled thyroid dysfunction
22. Subject has uncontrolled diabetes mellitus
23. Subject has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies) as determined by medical record review.
24. Subject has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected) as determined by medical record review.
25. Subject has received a live vaccine within 30 days prior to the first dose of trial treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2021-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tara Mitchell, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
Study already published

REFERENCES:
- [Result] Huang AC, Orlowski RJ, Xu X, Mick R, George SM, Yan PK, Manne S, Kraya AA, Wubbenhorst B, Dorfman L, D'Andrea K, Wenz BM, Liu S, Chilukuri L, Kozlov A, Carberry M, Giles L, Kier MW, Quagliarello F, McGettigan S, Kreider K, Annamalai L, Zhao Q, Mogg R, Xu W, Blumenschein WM, Yearley JH, Linette GP, Amaravadi RK, Schuchter LM, Herati RS, Bengsch B, Nathanson KL, Farwell MD, Karakousis GC, Wherry EJ, Mitchell TC. A single dose of neoadjuvant PD-1 blockade predicts clinical outcomes in resectable melanoma. Nat Med. 2019 Mar;25(3):454-461. doi: 10.1038/s41591-019-0357-y. Epub 2019 Feb 25. PMID 30804515
- [Derived] Sharon CE, Tortorello GN, Ma KL, Huang AC, Xu X, Giles LR, McGettigan S, Kreider K, Schuchter LM, Mathew AJ, Amaravadi RK, Gimotty PA, Miura JT, Karakousis GC, Mitchell TC. Long-term outcomes to neoadjuvant pembrolizumab based on pathological response for patients with resectable stage III/IV cutaneous melanoma. Ann Oncol. 2023 Sep;34(9):806-812. doi: 10.1016/j.annonc.2023.06.006. Epub 2023 Jul 4. PMID 37414215
- See also: Pubmed link — https://www.ncbi.nlm.nih.gov/pubmed/30804515

RESULTS

PARTICIPANT FLOW:
Groups:
- Neo-adjuvant/Adjuvant Pembrolizumab 200mgIV: Pembrolizumab 200 mg: Subjects received 1 dose of neoadjuvant pembrolizumab, followed by complete resection, and then a year of adjuvant pembrolizumab.
Period: Overall Study
Arm/Group | Neo-adjuvant/Adjuvant Pembrolizumab 200mgIV
Started | 33 (Consented)
Post Consent Screening | 30
Completed | 30
Not Completed | 3
Not completed — screen fail | 3

BASELINE CHARACTERISTICS:
Population: Subjects who were consented and completed post-consent screening
Groups:
- Neo-adjuvant/Adjuvant Pembrolizumab 200mg IV: Pembrolizumab 200 mg: Subjects received 1 dose of neoadjuvant pembrolizumab, followed by complete resection, and then a year of adjuvant pembrolizumab.
Arm/Group | Neo-adjuvant/Adjuvant Pembrolizumab 200mg IV
Number analyzed (Participants) | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 17
  >=65 years | 13
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 30
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 30
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 30
Stage at Study Entry [Number; unit: participants] — Stage IIIB (at least 1 bulky regional lymph node), IIIC (bulky regional lymph nodes and/or ulcerated primary tumor), Stage IV (distant metastasis)
  participants
    Stage IIIB | 12
    Stage IIIC | 17
    Stage IV | 1
Baseline LDH [Number; unit: participants]
  Normal | 30
  Elevated | 29
  No Data | 1
Primary Site [Number; unit: participants]
  cutaneous | 24
  unknown | 6
BRAF V600 [Number; unit: participants]
  Wild Type | 9
  Mutant | 7
  Unknown | 14
Prior Therapy [Number; unit: participants]
  PLX4032 | 1
  None | 29

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants (%) With CTCAE Graded Adverse Events
Description: Safety as defined by 1) all grade 3/4 adverse events and 2) any grade adverse event that occurred in>5% of patients. Toxicities are graded using CTCAE Version 4.
Time Frame: within 30 days of final study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Neo-adjuvant/Adjuvant Pembrolizaumab 200 mg IV
Number analyzed (Participants) | 30
Participants | 6

ADVERSE EVENTS:
Time Frame: 15 months
Description: All SAEs are reported. Grade 3-5 AEs and SAEs and occurring in at least 5% of subjects are reported.
Arm/Group | Neo-adjuvant/Adjuvant Pembrolizumab 200mg IV
All-Cause Mortality (participants affected / at risk) | 6/30
Serious Adverse Events (participants affected / at risk) | 6/30
Other Adverse Events (participants affected / at risk) | 2/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neo-adjuvant/Adjuvant Pembrolizumab 200mg IV (N=30)
Anaphylaxis (Immune system disorders) | 1 (1) — Grade 3 possibly related
esophageal obstruction (Gastrointestinal disorders) | 1 (1) — Grade 3 unrelated
colitis (Gastrointestinal disorders) | 1 (1) — Grade 3 unrelated
Enteritis (Immune system disorders) | 1 (1) — grade 3 enteritis possibly related
wound infection (Infections and infestations) | 1 (1) — grade 3 unrelated
sepsis (Infections and infestations) | 1 (2) — grade 4 unrelated
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neo-adjuvant/Adjuvant Pembrolizumab 200mg IV (N=30)
Rash (Skin and subcutaneous tissue disorders) | 2 (3) — Grade 3 rash

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-06-18): https://cdn.clinicaltrials.gov/large-docs/54/NCT02434354/Prot_SAP_000.pdf